CLINICAL TRIAL: NCT00111384
Title: Variation in Gene Expression in Neurofibromatosis Type 1
Brief Title: Study of Disease Severity in Adults With Neurofibromatosis Type 1 (NF1)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050152; 05-C-0152
Record Dates: First submitted 2005-05-19; First posted 2005-05-20 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-05-15

CONDITIONS: Neurofibromatosis Type 1; Legius Syndrome
Keywords: Phenotype; NF1-associated tumors; NF1; EQTL; Modifier Genes; Natural History; Neurofibroma; Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1; Legius syndrome; Neurofibroma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Affected participants, must have a correct clinical diagnosis of NF1.
- Group B: Unaffected individuals greater than 2 years of age who are relatives of participants.

SUMMARY:
This study may identify genes that predict the seriousness of neurofibromatosis type 1 (NF1). Finding these genes may explain why some people with NF1 have more medical problems than others. The study will also examine medical problems in NF1 that are rarely seen and are not well understood.

Male and female patients with NF1 who have gone through puberty may be eligible for this study, as well as patients of any age who have unique or under-recognized disease features. Affected and unaffected family members, including parents, siblings, and more distant relatives, may also be enrolled. Candidates are screened with a discussion of medical history or review of medical records, or both. Participants undergo the following procedures:

Patients with NF1

* Physical examination and family history
* Photographs of the iris of each eye
* Photographs of the back, abdomen and thigh to count skin tumors
* Photographs of the face and body (with underwear on) to help track growth and appearance
* Magnetic resonance imaging (MRI) of the spine (This test uses a magnetic field and radio waves to look for tumors and curvature of the spine. The patient lies still in the scanner, a narrow cylindrical device, wearing earplugs to muffle loud knocking sounds that occur during the scan. A contrast material called gadolinium is injected into a vein through a catheter to enhance the images.)
* Blood draw for genetic studies
* Possibly a skin biopsy (with the use of numbing medicine, removal of a small sample of skin tissue) to grow cells in the laboratory

Patients with NF1 who have unique or under-recognized disease features

* Physical examination and family history
* Blood draw for genetic studies
* Possibly a skin biopsy
* Possibly additional tests, such as blood work, x-rays, photographs, MRIs, ultrasounds, or other tests

Unaffected family members

* Blood draw for genetic studies
* Brief skin and eye examinations
* Possibly a skin biopsy for cell culture

Families are asked to give permission for researchers to recontact them for follow-up information, additional blood samples, or follow-up visit.

...

DETAILED DESCRIPTION:
We hypothesize that normal germline variation in gene expression accounts, in part, for variation in the clinical severity and phenotype of the monogenic disorder neurofibromatosis type 1 (NF1). The phenotype of NF1 is constituted by a variety of quantifiable features; we term these features sub-phenotypes . Our main focus is on sub-phenotypes with published evidence of variation in expression from an inherited component. These include our primary sub-phenotype of spinal neurofibroma burden (quantified by MRI of spinal neurofibromas) and the secondary sub-phenotypes of dermal neurofibroma burden, head circumference, number of Lisch nodules, scoliosis, history of plexiform neurofibromas, and height. Other sub-phenotypes, as collected by a routine history and physical, will also be evaluated.

According to our hypothesis, the severity of a sub-phenotype will correlate with heritable differences in the germline expression of certain genes. As an example, consider a spectrum of individuals affected with the primary sub-phenotype of spinal neurofibroma burden. For most genes, there will be no relationship of expression level to the number of spinal neurofibromas. However, some genes will have a direct (or inverse, or other) correlation of their level of expression and the number of neurofibromas. Such genes would be considered as candidate modifier genes. The secondary sub-phenotypes will also be analyzed in a similar way. To limit false positives, candidate genes will then be tested for association (using the transmission/disequilibrium test, TDT) with the appropriate sub-phenotype.

Recruitment will be focused on identifying individuals with a range of severity of the primary sub-phenotype, spinal neurofibroma burden. We will primarily recruit post-pubertal individuals who meet the 1988 NIH criteria for neurofibromatosis type 1 (NIH Consensus Development Conference 1988). We will exclude those with recognized segmental or mosaic NF1. The rate of cutaneous neurofibroma growth and number is known to vary widely; these tumors typically appear in adolescence. For this reason we will ascertain patients after puberty. We expect most individuals to be 18 years or older, but will also accept post-pubertal pediatric patients (and use a hand film to demonstrate bone age). Parents (whether affected or not) are critical when using family-based tests of association (like the TDT) and tests of linkage and will also be recruited.

Tests of association with the TDT require trios (mother, father, proband). Multiple trios can be derived from a single family, if there are multiple affected individuals within the family. We set a recruitment goal of 100 trios and a ceiling of 1500 individuals (500 affected individuals, plus 1000 parents or additional sibs in about 400 families).

In the interest of improving care for people living with NF1, this protocol also seeks to characterize, at the PI s discretion, individuals with unique or under-recognized features of NF1 as well as individuals with NF1-like phenotypes, including those patients with a known or suspected RAS pathway disorder.

ELIGIBILITY:
* INCLUSION CRITERIA:

Group A: All affected individuals in a family who are post-pubertal male and female individuals and who meet the 1988 NIH criteria for neurofibromatosis type 1 (NIH Consensus Development Conference 1988).

Group B: Unaffected individuals greater than 2 years of age who are relatives of participants (especially parents, but also siblings) are eligible to enroll and are critical to the success of the study. These individuals may be of any gender and ethnicity. If the individual is pre-pubertal, s/he must have a brief evaluation at the NIH Clinical Center (abbreviated medical history and skin and eye exam) to ensure s/he is not affected with NF1.

Group C: individuals with unique or under-recognized features of NF1 of any age, gender or ethnicity and must have a correct clinical diagnosis of NF1 (NIH Consensus Development Conference 1988). all Group C participants enrolling in the study identify a physician who will be responsible for follow-up care so this can be arranged (if needed) at the conclusion of the evaluation at NIH.

For healthy normal volunteers used for MRI imaging of the spine, we will aim to recruit one male and one female from each of 5 decades (18-30 years, 31-40 years, 41-50 years, 51-60 years, 61-70 years). These individuals may be of any ethnicity.

Additional requirements include:

1. If female and of child-bearing age, must be willing to have a serum pregnancy test (HCG) and
2. Willingness to undergo a brief, focused history and physical exam to rule out occult spine pathology and to verify there are no contra-indications to spinal MRI imaging.

EXCLUSION CRITERIA:

EXCLUSION CRITERIA FOR GROUP A INDIVIDUALS INCLUDE:

1. Any history of administration (or current use) of radiation therapy, chemotherapeutic agents or biologic agents (experimental or not) that resulted in a documented significant change in spinal neurofibroma tumor burden or growth.
2. Any history of administration (or current use) of medication that might reasonably be expected to alter the natural history of tumor growth (examples include pirfenidone, interferon, farnesyl transferase inhibitor (FTI), MTX/VBL, thalidomide, growth hormone) or cause significant changes in gene expression profile.
3. Any history of surgery to significantly debulk spinal neurofibromas
4. Pregnancy/Lactation. If an affected pregnant or lactating woman is eligible for participation, we will request that she enroll after the conclusion of the pregnancy or lactation.
5. Cognitive delay in an adult or minor to the extent that sedation is required to obtain MRI.
6. Presence or suspected presence of hardware (Harrington rods) or metallic objects (e.g. shrapnel, aneurysm clips) or history of exposure to such objects (e.g. welding) that preclude MRI imaging.
7. Inability or unwillingness to tolerate a 1-hour (or more) MRI protocol.
8. Patients will be excluded if they cannot travel to the NIH because of their medical condition OR are less than 2 years of age. The PI may decline to enroll a patient for other reasons.

EXCLUSION CRITERIA FOR GROUP B INDIVIDUALS INCLUDE:

1) A non-affected pregnant or lactating woman in a family for whom LCL immortalization will not be performed may participate. However, if she is a member of a multi-affected family (and thus her blood will be used to prepare LCLs) we will request that she donate a blood sample at the conclusion of her pregnancy or upon the weaning of her child.

EXCLUSION CRITERIA FOR GROUP C INDIVIDUALS INCLUDE:

1) Less than 2 years of age.

EXCLUSION CRITERIA FOR HEALTHY, NORMAL VOLUNTEERS INCLUDE:

1. Pregnancy or lactation (a serum HCG level will be drawn on all child-bearing age women). Women unwilling to have a serum pregnancy test cannot participate.
2. Any history of spine surgery or significant spinal disease (severe arthritis, autoimmune disorders, severe scoliosis, kyphosis or lordosis, cancer, NF1, NF2, or schwannomatosis)
3. Any active spine-related complaints: e.g. persistent back pain, radicular symptoms
4. Clinically significant medical condition that, in the opinion of the investigator, would compromise the patient's safety or affect his/her MRI (e.g., diabetes mellitus, chronic hypertension, severe anemia, kidney disease, heart disease [angina, arrhythmias, congestive heart failure]).
5. Previous eye surgery of any kind.
6. Inability to provide informed consent.
7. Permanent tattooed makeup (eyeliner, lip, etc) or general tattoos. Subjects with tattoos will be excluded if those are in a dangerous location in the body or made with colors (e.g. dark blue and dark green) whose content in iron cannot be definitely ruled out by the Investigators.
8. Any non-organic implant or any other device such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitro, hormones) that may cause problems if removed even temporarily, any metallic implants or objects, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunt.
9. Cerebral or other aneurysm clips.
10. Shrapnel or other metal imbedded in the subject's body (such as from war wounds or accidents).
11. Previous work in metal fields or with machines that may have left any metallic fragments in or near the subject's eyes.
12. A severe auto accident in the past so if it is uncertain whether any metal may still be imbedded in the subject's body.
13. Any psychological contraindications for MRI (e.g., suffer from claustrophobia). This will be assessed at the time when the medical history will be collected.
14. Any contraindications to having study procedures done.
15. Dental work such as crowns or bridges with indeterminate metals
16. The PI may decline to enroll a patient for other reasons.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with the genetic disorder Neurofibromatosis Type 1
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2005-07-27 (Actual)

PRIMARY OUTCOMES:
Phenotype individuals and family members affected with NFl by routine history and physical. | ongoing
  Phenotype severityPhenotype individuals and family members affected with NF1 by routine history and physical. The primary (spinal neurofibroma burden) and secondary (dermal neurofibroma burden, head circumference, number of Lisch nodules, scoliosis, history of plexiform neurofibromas, height) sub- phenotypes will be quantified with as appropriate technology (MRI, iris exam and photography, physical exam, medical history).
Identify candidate modifier genes by determining the correlation coefficient of the level of gene expression and the severity of each sub- phenotype (as phenotyped in Aim 1). | ongoing
  Identify candidate modifier genes by determining the correlation coefficient of the level of gene expression and the severity of each sub- phenotype (as phenotyped in Aim 1).
Characterize individuals with 1) unique or under-recognized features of NFl, and 2) individuals with NFl-like phenotypes, including those patients with a known or suspected RAS pathway disorder. | ongoing
  Characterize individuals with 1) unique or under-recognized features of NFl, and 2) individuals with NFl-like phenotypes, including those patients with a known or suspected RAS pathway disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Stewart, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical data will be shared with collaborators under appropriate agreements.
Supporting Information: Study Protocol
Time Frame: At the time of a request and as long as needed.
Access Criteria: De-identified clinical data will be shared with collaborators under appropriate agreements.

REFERENCES:
- [Background] Pemov A, Park C, Reilly KM, Stewart DR. Evidence of perturbations of cell cycle and DNA repair pathways as a consequence of human and murine NF1-haploinsufficiency. BMC Genomics. 2010 Mar 22;11:194. doi: 10.1186/1471-2164-11-194. PMID 20307317
- [Background] Stewart DR, Brems H, Gomes AG, Ruppert SL, Callens T, Williams J, Claes K, Bober MB, Hachen R, Kaban LB, Li H, Lin A, McDonald M, Melancon S, Ortenberg J, Radtke HB, Samson I, Saul RA, Shen J, Siqveland E, Toler TL, van Maarle M, Wallace M, Williams M, Legius E, Messiaen L. Jaffe-Campanacci syndrome, revisited: detailed clinical and molecular analyses determine whether patients have neurofibromatosis type 1, coincidental manifestations, or a distinct disorder. Genet Med. 2014 Jun;16(6):448-59. doi: 10.1038/gim.2013.163. Epub 2013 Nov 14. PMID 24232412
- [Background] Brems H, Park C, Maertens O, Pemov A, Messiaen L, Upadhyaya M, Claes K, Beert E, Peeters K, Mautner V, Sloan JL, Yao L, Lee CC, Sciot R, De Smet L, Legius E, Stewart DR. Glomus tumors in neurofibromatosis type 1: genetic, functional, and clinical evidence of a novel association. Cancer Res. 2009 Sep 15;69(18):7393-401. doi: 10.1158/0008-5472.CAN-09-1752. Epub 2009 Sep 8. PMID 19738042
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-C-0152.html